CLINICAL TRIAL: NCT04007380
Title: Psychosocial, Cognitive, and Behavioral Consequences of Sleep-disordered Breathing in Spinal Cord Injured People
Brief Title: Psychosocial, Cognitive, and Behavioral Consequences of Sleep-disordered Breathing After SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-5072
Record Dates: First submitted 2019-03-25; First posted 2019-07-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries; Sleep Apnea
Keywords: Spinal cord injuries; Sleep-related breathing disorders
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPAP-therapy arm (Other): This single-arm clinical trial will examine the effects of 4-month period CPAP therapy in individuals living with SCI. The CPAP will be adjusted according to the results of the auto-titrating CPAP testing for each participant.
  Interventions: Other: Continuous positive airway pressure (CPAP) therapy

INTERVENTIONS:
Other: Continuous positive airway pressure (CPAP) therapy — The participants will undergo CPAP therapy for 4 consecutive months in the management of moderate-to-severe SRBDs

SUMMARY:
This clinical trial will examine the efficacy of continuous positive airway pressure (CPAP) therapy in improving psychosocial, neurocognitive and behavioral consequences of moderate-to-severe sleep-related breathing disorders (SRBDs) in people living with spinal cord injury (SCI).

DETAILED DESCRIPTION:
SCI is a potentially catastrophic event for individuals who may sustain motor, sensory, and autonomic deficit, as well as secondary conditions including SRBDs. The SRBDs include central, obstructive and mixed sleep apnea that can occur in up to 50% of the paraplegics and up to 91% of the motor complete tetraplegics. Although the frequency of SRBDs after SCI is much greater than in able-bodied people, this condition is still a largely under-recognized in the SCI population.

With this, the investigators hypothesize that regular use of CPAP for treatment of moderate-to-severe SRBDs in individuals living with SCI significantly improve their fatigue, depressive symptoms, anxiety, cognitive impairment, quality of life, and social and work participation. This research project will include: (i) a single-arm clinical trial to evaluate the efficacy of nightly use of CPAP for 4 consecutive months in the management of moderate-to-severe SRBDs among 24 adults with subacute to chronic, cervical or thoracic, complete or incomplete SCI; and (ii) a qualitative study of the challenges experienced by the 24 people with SCI who undergo an unattended-hospital or home-based sleep study for diagnosis of SRBDs followed by CPAP therapy.

Overall, this clinical study has the potential to ultimately improve fatigue, mood, cognition, quality of life, and social and work participation of people living with SCI, by examining under-explored links with the SRBDs.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults 18 years of age or older
* Have traumatic cervical/thoracic (injury level at C5 to T10), severe or moderate (AIS A, B, or C) SCI who were not diagnosed with a sleep disorder prior to the injury.
* At least 2 months after injury
* Clinical warning symptoms and/or signs for SRBDs

Exclusion Criteria:

* Patients with a non-traumatic spinal cord disease at risk for neurologic progression
* Concomitant diseases of the central nervous system
* Preinjury chronic pain
* Psychiatric disorders that may prevent the participant to be compliant to the study protocol requirements
* Neuromuscular diseases
* Current substance misuse
* History of primary hypersomnia
* Hypothyroidism
* Moderate or severe iron deficiency anemia
* Active infection
* Kidney failure
* Epilepsy
* Chronic fatigue syndrome
* Vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Change in Fatigue Severity Scale from baseline to after 4-month period of CPAP therapy
  Self-reported (or administered by an interviewer) scale where participants choose one of seven levels of agreement for each question. Range from 9 (best outcome) to 63 (worst outcome). The primary outcome is the difference between post-intervention and pre-intervention Fatigue Severity Scales.

SECONDARY OUTCOMES:
Epworth Sleepiness Score | Change in Epworth Sleepiness Score from baseline to after 4-month period of CPAP therapy
  Self-reported (or administered by an interviewer) where participants answer the 8 brief questions. Range from 0 (best outcome) to 24 (worst outcome). This secondary outcome comprises the difference between post-intervention and pre-intervention Epworth sleepiness scores.
Medical Outcomes Study Sleep Scale | Change in Medical Outcomes Study Sleep Scale from baseline to after 4-month period of CPAP therapy
  Self-reported scale that consists of 12 Likert-type items assessing six dimensions of sleep problems: sleep disturbance (i.e. difficulty initiating or maintaining sleep), snoring, respiratory problems, sleep quantity, sleep adequacy, and daytime somnolence). Higher scores for the domains of sleep disturbance, somnolence and sleep indices indicate worse sleep disturbances, whereas lower scores for sleep quantity and sleep adequacy indicate worse sleep disturbances.
Depression, Anxiety & Stress Scales- 21 | Change in Depression, Anxiety & Stress Scales- 21 from baseline to after 4-month period of CPAP therapy
  Self-reported (or administered by an interviewer) scale where participants rate questions on depression, anxiety and stress. Depression subscale varies from 0 (best outcome) to 21 (worst outcome). Anxiety subscale varies from 0 (best outcome) to 21 (worst outcome). Stress subscale varies from 0 (best outcome) to 21 (worst outcome). This secondary outcome comprises the difference in the overall pre-intervention and post-intervention DASS-21 scores.
Montreal Cognitive Assessment (MoCA) test | Change in Montreal Cognitive Assessment (MoCA) score from baseline to after 4-month period of CPAP therapy
  Cognitive test administered by an interviewer.

OTHER OUTCOMES:
Face-to-face, 1-hour interview for qualitative analysis | At completion of the 4-month period of CPAP therapy
  Qualitative study of the challenges experienced by the 24 people with SCI who undergo an unattended-hospital or home-based sleep study for diagnosis of SRBDs followed by CPAP therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Furlan, MD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Lyndhurst Centre, KITE - TRI UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No